CLINICAL TRIAL: NCT04504565
Title: The Efficacy of 99mTc-3PRGD2 SPECT/CT Imaging in the Diagnosis of Lymph Node Metastasis of Esophageal Carcinoma
Brief Title: 99m Tc-3PRGD2 SPECT/CT Imaging in the Diagnosis of Lymph Node Metastasis of Esophageal Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MIC-ESO-003
Record Dates: First submitted 2020-07-29; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Esophageal Cancer; Lymph Node Metastases; Diagnoses Disease
MeSH Terms: conditions — Esophageal Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 99mTc-3PRGD2 (Experimental): intravenous injection of 0.3 mCi/kg of 99mTC-3PRGD2, patients underwent single-photon emission computed tomography/COMPUTED tomography (SPECT/CT) examination.
  Interventions: Diagnostic Test: 99mTc-3PRGD2

INTERVENTIONS:
Diagnostic Test: 99mTc-3PRGD2 — intravenous injection of 0.3 mCi/kg of 99mTc-3PRGD2

SUMMARY:
The esophageal squamous cell carcinoma (ESCC) has high prevalence and mortality in China, which become a severe challenge for public health. The molecular imaging technology has been developed for visualization and precise diagnosis of the tumors. Integrin αvβ3 is a specific marker for tumor. Noninvasive visualization and quantitative analysis of integrin αvβ3 expression provide new opportunities for tumor diagnosis, identification and efficacy monitoring. The peptide containing Arg-Gly-Asp (RGD) can specifically bind to integrin αvβ3 receptor with high selectivity and affinity to achieve the detecting tumor .The SPECT/CT with 99mTc-3PRGD2 has a high specificity in the diagnosis of mediastinal lymphnode metastasis and a greater value in the decision-making of lymphnode dissection.

This study is a single-center self-controlled study, It is planned to enroll 30 patients with esophageal cancer , preliminarily confirmed by endoscopic biopsy, . After intravenous injection of 0.3 mCi/kg of 99mTC-3PRGD2, patients underwent single-photon emission computed tomography/computed tomography (SPECT/CT) examination.Subsequently, the patients received chest/abdomen enhanced CT and 18F fluorodeoxyglucose (18F-FDG) positron emission computed tomography /CT (PET/CT) for diagnosis. According to the determination of the researcher, patients who were suitable for surgery received surgery to obtain surgical pathology; For patients who were not suitable for surgery, ultrasound-guided lyphnode biop was performed .In this study, pathological specimens were obtained from gastroscopy, surgical pathology, or ultrasound-guided lymph node biopsy. The diagnostic accuracy, sensitivity , specificity and safety of SPECT/CT with 99mTc-3PRGD2 were evaluated and compared with PET-CT and enhanced CT.

DETAILED DESCRIPTION:
Screening period All patients will be during the screening screening assessment, specific include: the signing of the ICF, demographic data, drug allergy history and history, height, weight, physical examination, vital signs, electrocardiogram (ECG) examination, laboratory examination, blood pregnancy test records (if applicable), endoscopic biopsy, AE and drug combination, check into/standard. Qualified patients will enter the administration period after screening and confirmation. Administration period (from Administration to safety follow-up) day of administration (study day 1): before administration of the experimental drug, 12-lead ECG, laboratory test (fasting) and vital signs were measured. Subsequently, the experimental drug was injected intravenously at 0.3 ± 20% mCi/kg, and subjects underwent urination and SPECT/CT examination 40 min after administration. AE and combined medication were recorded. The next day after administration (day 2 of the study): 12-lead ECG, laboratory examination (fasting), vital signs were measured, AE and combined medication were recorded. Between the administration of 99mTc-3PRGD2 and the safety follow-up, the investigator determined that chest/abdomen enhanced CT and PET/CT were performed at an optional date.

Safety follow-up (day 14±2 of the study or before the next clinical intervention, whichever is shorter) :

12 lead ECG, laboratory test (fasting), measurement of vital signs, blood pregnancy (women of childbearing age only), AE and combined medication were recorded.Lymph node histopathology was obtained by surgery in patients suitable for surgery, and by ultrasound-guided lymph node biopsy in patients unsuitable for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Esophageal cancer was confirmed by Endoscopic biopsy
* Clinical laboratory tests (heart, liver, kidney, blood) and other indicators are in the normal range, or the abnormalities have no clinical significance (NCS), or the abnormalities have clinical significance (CS) but do not affect the implementation of surgery or lymph node puncture;
* The patient being able to follow scheduled visits, treatment plans and laboratory tests.

Exclusion Criteria:

* Female patients who plan to become pregnant within 6 months, or are pregnant or breastfeeding;
* Allergic to test drugs, allergic constitution or multiple drugs;
* Weight over 100 kg;
* Claustrophobia;
* Cannot tolerate both arms raised and supine for 15-30 minutes;
* The investigator considers it inappropriate to participate in this clinical trial;
* The patient participated in or participating in other clinical trials within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
the accuracy of SPECT/CT with 99mTc-3PRGD2 in the diagnosis of lymph node metastasis | 14 days
  To evaluate the accuracy of SPECT/CT with 99mTc-3PRGD2 in the diagnosis of lymph node metastasis of esophageal carcinoma，according to the pathological analysis, according to the pathological analysis.
the sensitivity of SPECT/CT with 99mTc-3PRGD2 in the diagnosis of lymph node metastasis | 14 days
  To evaluate the sensitivity of SPECT/CT with 99mTc-3PRGD2 in the diagnosis of lymph node metastasis of esophageal carcinoma，according to the pathological analysis, compared with PET-CT and enhanced CT.

SECONDARY OUTCOMES:
The Incidence of Adverse Events | 14 days
  To evaluate the safety of 99mTc-3PRGD2 in SPECT/CT in the diagnosis of lymph node metastasis of esophageal carcinoma

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang Z, Zhao X, Ding C, Wang J, Zhang J, Wang F. (99m)Tc-3PRGD2 SPECT/CT Imaging for Monitoring Early Response of EGFR-TKIs Therapy in Patients with Advanced-Stage Lung Adenocarcinoma. Cancer Biother Radiopharm. 2016 Sep;31(7):238-45. doi: 10.1089/cbr.2016.2052. Epub 2016 Aug 26. PMID 27563805
- [Result] Jin X, Liang N, Wang M, Meng Y, Jia B, Shi X, Li S, Luo J, Luo Y, Cui Q, Zheng K, Liu Z, Shi J, Li F, Wang F, Zhu Z. Integrin Imaging with 99mTc-3PRGD2 SPECT/CT Shows High Specificity in the Diagnosis of Lymph Node Metastasis from Non-Small Cell Lung Cancer. Radiology. 2016 Dec;281(3):958-966. doi: 10.1148/radiol.2016150813. Epub 2016 Jul 29. PMID 27479638
- [Result] Ji B, Chen B, Wang T, Song Y, Chen M, Ji T, Wang X, Gao S, Ma Q. (9)(9)mTc-3PRGD(2) SPECT to monitor early response to neoadjuvant chemotherapy in stage II and III breast cancer. Eur J Nucl Med Mol Imaging. 2015 Aug;42(9):1362-70. doi: 10.1007/s00259-015-3062-1. Epub 2015 May 7. PMID 25947573
- [Result] Ma Q, Min K, Wang T, Chen B, Wen Q, Wang F, Ji T, Gao S. (99m)Tc-3PRGD 2 SPECT/CT predicts the outcome of advanced nonsquamous non-small cell lung cancer receiving chemoradiotherapy plus bevacizumab. Ann Nucl Med. 2015 Jul;29(6):519-27. doi: 10.1007/s12149-015-0975-5. Epub 2015 Apr 25. PMID 25911312
- [Result] Ma Q, Chen B, Gao S, Ji T, Wen Q, Song Y, Zhu L, Xu Z, Liu L. 99mTc-3P4-RGD2 scintimammography in the assessment of breast lesions: comparative study with 99mTc-MIBI. PLoS One. 2014 Sep 24;9(9):e108349. doi: 10.1371/journal.pone.0108349. eCollection 2014. PMID 25250628
- [Result] Liu L, Song Y, Gao S, Ji T, Zhang H, Ji B, Chen B, Jia B, Wang F, Xu Z, Ma Q. (99)mTc-3PRGD2 scintimammography in palpable and nonpalpable breast lesions. Mol Imaging. 2014;13(5). doi: 10.2310/7290.2014.00010. PMID 24825112
- [Result] Ma Q, Ji B, Jia B, Gao S, Ji T, Wang X, Han Z, Zhao G. Differential diagnosis of solitary pulmonary nodules using (9)(9)mTc-3P(4)-RGD(2) scintigraphy. Eur J Nucl Med Mol Imaging. 2011 Dec;38(12):2145-52. doi: 10.1007/s00259-011-1901-2. Epub 2011 Aug 27. PMID 21874323
- [Result] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342